CLINICAL TRIAL: NCT06835049
Title: Feasibility of Total Neoadjuvant Treatment With HYPErthermia in Patients With High-risk Extremity and Trunk Soft Tissue Sarcoma (TNT-HYPE). A Multicenter, Single Arm, Open Label, Phase II Trial
Brief Title: Feasibility of Total Neoadjuvant Treatment With HYPErthermia in Patients With High-risk Extremity and Trunk Soft Tissue Sarcoma (TNT-HYPE)
Acronym: TNT-HYPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 57/24
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma,Soft Tissue
Keywords: Sarcoma, soft-tissue; TNT-HYPE; phase II; Neoadjuvant Treatment; hyperthermia
MeSH Terms: conditions — Sarcoma; Hyperthermia | interventions — Doxorubicin; Ifosfamide; Dacarbazine; Diathermy; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Multicenter, single arm, open label, phase II trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Treatment (Experimental): Trial treatment consists of 3 neoadjuvant cycles of doxorubicin with either ifosfamide or dacarbazine (the latter only in case of leiomyosarcoma) combined with hyperthermia (HT), followed by radiotherapy (RT) and surgery. Each chemotherapy cycle will last 3 weeks. Trial treatment will last approximately 20 weeks. After surgery, a follow-up period of 36 months per patient is foreseen.
  Interventions: Drug: Doxorubicin; Drug: Ifosfamide; Drug: Dacarbazine; Other: Hyperthermia; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Doxorubicin — Trial treatment consists of 3 neoadjuvant cycles of doxorubicin with either ifosfamide or dacarbazine (the latter only in case of leiomyosarcoma). Doxorubicin will be given at a dose of 75 mg/m2 Body surface area (BSA) on day 1 of each cycle as a intravenous infusion over 15 minutes.
Drug: Ifosfamide — Trial treatment consists of 3 neoadjuvant cycles of doxorubicin with either ifosfamide or dacarbazine (the latter only in case of leiomyosarcoma). Ifosfamide will be given at a dose of 3 g/m2 BSA on days 1 to 3 of each cycle, for a total dose per cycle of 9 g/m2 BSA, as an intravenous infusion of 3 g/m2 daily over 4 hours.
Drug: Dacarbazine — Trial treatment consists of 3 neoadjuvant cycles of doxorubicin with either ifosfamide or dacarbazine (the latter only in case of leiomyosarcoma). Dacarbazine will be given at a daily dose of 300 mg/m2 BSA on days 1 to 3 of each cycle, for a total dose per cycle of 900 mg/m2 BSA, as an intravenous infusion over 30 minutes.
Other: Hyperthermia — Hyperthermia (HT) sessions are scheduled on days 1 and 3 of each chemotherapy cycle. The duration of the preheating phase is always 30 minutes. Together with the treatment phase of 60 minutes, the duration of a HT session is uniformly 90 minutes (Total treatment time). On days 2, chemotherapy will be applied without HT.
Radiation: Radiotherapy — Radiotherapy (RT) treatment should start ideally 19 days after last chemotherapy dose received (range -4 / +7), preferably on a Monday to omit that the last RT fractions will be applied directly after the weekend. Start of RT can be postponed up to 14 days due to medical reasons without violating treatment protocol.
  Patients will preferably receive normofractionated RT to a total dose of 50 Gy in 25 fractions of 2 Gy over 5 weeks23.
  Alternatively, patients can receive a moderate hypofractionated RT to either a total dose of 42.75 Gy in 15 fractions of 2.85 Gy over 3 weeks or a total dose of 42 Gy in 14 fractions of 3 Gy over 2 weeks and four days41. The respective total treatment time changes respectively.
  The RT treatment should be delivered once daily except on weekends.
Procedure: Surgery — Standard of care surgical resection must be done by an experienced sarcoma surgeon. All lesions of the trunk and extremities will be resected after total neoadjuvant treatment with chemotherapy, HT and RT.
  Surgery will take place preferentially 6 weeks (+/- 2 weeks) after end of radiation.

SUMMARY:
Soft tissue sarcomas (STSs) are rare cancers with a 5-year survival rate of 60%, and there is no standard treatment for high-risk extremity and trunk STSs (eSTS). A phase III trial suggests that adding moderate regional hyperthermia (HT) to anthracycline-based chemotherapy, followed by surgery and radiotherapy (RT), can improve 10-year overall survival by 10%. This trial aims to optimize treatment by combining the most effective regimens from chemotherapy, HT, RT, and surgery, and will evaluate the feasibility of this new total neoadjuvant treatment (TNT) approach.

DETAILED DESCRIPTION:
Soft tissue sarcomas (STSs) are rare cancers with a 5-year survival rate of only 60%. There is no international standard treatment for high-risk extremity and trunk STSs (eSTS). Current evidence from a phase III trial suggests that adding moderate regional hyperthermia (HT) to anthracycline-based chemotherapy followed by surgery and radiotherapy (RT) can improve survival rates, showing a 10% improvement in 10-year overall survival.

The aim of this trial is to optimize the treatment for this high-risk group. To achieve this, the assumed most effective treatment regimens from each treatment modality (chemotherapy, HT, RT, and surgery) were identified and combined into an optimized treatment protocol. Neoadjuvant chemotherapy in this population is not yet broadly accepted as standard of care. Furthermore, this new total neoadjuvant treatment (TNT) approach has not yet been investigated prospectively and in addition, the patients have to get their HT treatment potentially in a hospital distant from their domicile. Therefore, we will evaluate in this trial the feasibility of this new treatment schedule as primary endpoint.

Trial treatment consists of 3 neoadjuvant cycles of doxorubicin with either ifosfamide or dacarbazine (the latter only in case of leiomyosarcoma) combined with HT, followed by RT and surgery. Each chemotherapy cycle will last 3 weeks. Trial treatment will last approximately 20 weeks. After surgery, a follow-up period of 36 months per patient is foreseen.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically confirmed primary high-risk Soft tissue sarcoma (STS) of extremity or trunk.
* High-risk according to the prognostic Sarculator tool: 10-year OS probability < 60%5.
* Resectable tumor: resectability is based on pre-operative imaging and has to be defined by the local treating sarcoma team. A patient is not considered resectable when the expectation is that only a R2 resection is feasible.
* Measurable disease per RECIST v1.1.
* Diagnostic biopsy is available for the central pathology review.
* Candidate for chemotherapy regimen according to protocol.
* Candidate for loco-regional HT.
* Adequate bone marrow function, hepatic function, renal function, cardiac function and coagulation function.

Main Exclusion Criteria:

* Metastatic disease.
* Previous Whoops resection.
* Ex-ulcerating tumors or tumors infiltrating the skin.
* Other invasive malignancy within 5 years, with the exception of adequately treated non melanoma skin cancer, localized cervical cancer, localized and Gleason ≤ 6 prostate cancer.
* Any previous radiotherapy (RT) or systemic therapy for the present tumor.
* Previous treatment with maximum cumulative doses (450 mg/m² doxorubicin or equivalent 900 mg/m² epirubicin) of doxorubicin, daunorubicin, epirubicin, idarubicin, and/or other anthracyclines and anthracenediones.
* Concomitant or recent (within 30 days of registration) treatment with any other experimental drug.
* Concomitant use of other anti-cancer drugs or RT.
* No metal implants in the region of tumor or cardiac implant electronic devices (CIEDs).
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last 12 months, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia), significant QT-prolongation, uncontrolled hypertension.
* Active and uncontrolled infections, in particular urinary tract infections.
* Inflammation of the urinary bladder (interstitial cystitis).
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to registration.
* Vaccination with live vaccines within 30 days prior to registration.
* Known hypersensitivity to trial drug(s) or to any component of the trial drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Protocol feasibility rate | End of treatment approx. 20 weeks after registration
  PFR defined as percentage of patients who are able to finish the following planned trial treatment parts according to protocol

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From the date of registration until the date of local or distant relapse, progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 3 years after registration
  DFS defined as
  * time from registration until local or distant relapse,
  * or, if tumor has not been operated, time from registration until progression according to RECIST v1.1,
  * or death from any cause, whichever occurs first.

OTHER OUTCOMES:
Objective response rate (ORR) | From the date of registration until the date of progressive disease according to RECIST v1.1 or death, whichever occurs first, assessed up to 3 years after registration
  ORR assessed by the independent response reviewer and defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 during trial treatment and before surgery.
Pathologic complete response (pCR) | End of treatment approx. 20 weeks after registration
  pCR rate, assessed by the central pathologist and defined as proportion of patients with ≤ 10% viable cells (equivalent to EORTC-STBSG response grade A-C43) in the resection specimen. pCR rate will be evaluated in resected patients only.

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Stutz, MD, Study Director — Insel Gruppe AG, University Hospital Bern; Attila Kollàr, MD, Study Chair — University of Bern
Locations (8):
- Switzerland (8):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital Basel, Basel
  - EOC - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Inselspital Bern - Universitätsklinik für Radioonkologie, Bern
  - CHUV - Swiss Cancer Center Lausanne, Lausanne
  - hoch Health Ostschweiz - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Universitätsspital Zürich, Zurich